CLINICAL TRIAL: NCT04653493
Title: Phase I Clinical Trial Evaluating Safety of CD19 CAR-T Cells in Patients With Relapsed or Refractory Acute B-cell Lymphoblastic Leukemia (R/R B-ALL)
Brief Title: CD19 Targeted CAR T Cell Therapy in Patients With Relapsed/ Refractory B Cell Acute Lymphoblastic Leukaemia (ALL)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sabz Biomedicals (Industry)
Collaborators: Gene Therapy Research Center, Shariati Hospital, Tehran University of Medical Sciences, Iran (Unknown); Research Institute for Oncology- Hematology and Cell Therapy (RIOHCT), Tehran University of Medical Sciences, Iran (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19 CAR T Cells for R/R ALL
Record Dates: First submitted 2020-11-22; First posted 2020-12-04 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Relapsed B Cell Acute Lymphoblastic Leukemia (ALL); Refractory B Cell Acute Lymphoblastic Leukemia (ALL)
Keywords: CD19+ B-cell Acute Lymphoblastic Leukemia; CAR T cell; Relapsed/Refractory B cell acute lymphoblastic leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; fludarabine; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR-T cells (Experimental): Pediatric or adolescent/young adult patients with CD19+ relapsed or refractory B cell acute lymphoblastic leukemia (R/R B-ALL)
  Interventions: Biological: CD19 CAR engineered autologous T-cells; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna

INTERVENTIONS:
Biological: CD19 CAR engineered autologous T-cells — Given IV
  Following preconditioning with lymphodepleting chemotherapy (cyclophosphamide and fludarabine) patients will be treated with CD19 Chimeric Antigen Receptor (CAR) T cells as a single or split dose (day 0, 1 and 2, CAR cells will be intravenously infused at the 10%, 30% and 60% ratio respectively). Dosing of CD19 CAR-T cells will follow a dose-escalation schema, with dose changes based on dose-limiting toxicities.
Drug: Cyclophosphamide — Given IV
Drug: Fludarabine — Given IV
Drug: Mesna — Given IV

SUMMARY:
This is a single-arm, open-label, phase I study (safety and dose escalation) of autologous Chimeric Antigen Receptor (CAR) T-cells targeting CD19 in patients with relapsed/refractory B cell acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
In this single-center, open-label, nonrandomized, no control, prospective clinical trial, pediatric or adolescent/young adult patients with CD19+ relapsed or refractory B cell acute lymphoblastic leukemia (R/R B-ALL) will be enrolled.

Eligible patients will receive CAR T product intravenously as a single or split dose following pre-conditioning by a lymphodepleting chemotherapeutic regimen and will then enter a 30-day follow-up period to monitor adverse events using the NCI CTCAE (version 5.0).

ELIGIBILITY:
Inclusion Criteria:

CD19+ ALL patients with any of the following:

1. Relapsed or Refractory CD19 positive B-cell acute lymphoblastic leukemia (R/R B-ALL) A. Primary refractory disease despite at least 2 cycles of an intensive chemotherapy regimen designed to induce remission B. Refractory disease despite salvage therapy C. 2nd or greater relapse D. Any relapse after allogeneic hematopoietic stem cell transplantation
2. Informed consent explained to and signed by patient/parents or legal guardian.
3. The Karnofsky (age ≥10 years)/Lansky (age <10 years) performance status score over 50 points.
4. Expected to survive for more than 3 months.
5. Patients with a history of prior allogeneic hematopoietic stem cell transplant (HSCT) must be at least 3 months from HSCT at the time of CD19 CAR-T cells infusion and also have not received a donor lymphocyte infusion (DLI) within the 28 days prior to apheresis.
6. Important organ function is satisfied: Heart ultrasound indicates cardiac ejection fraction ≥ 50%, no obvious abnormality in ECG; Adequate pulmonary function defined as forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry ≥ 92% on room air if the patient is unable to perform pulmonary function testing; creatinine clearance calculated by Cockcroft-Gault formula ≥ 50 ml/min/1.73m2; Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age; Total Bilirubin ≤ 3 times the upper limit of normal for age.
7. Absolute lymphocyte count ≥ 0.5 x 10⁹/L.
8. Hemoglobin ≥ 8 g/dl (can be transfused).
9. Platelet count ≥ 20,000/μL (can be transfused).
10. Meets eligibility criteria to undergo autologous apheresis.

Exclusion Criteria:

1. Isolated extra-medullary disease relapse.
2. Active CNS involvement of ALL (CNS Grade 3 per National Comprehensive Cancer Network guidelines).
3. Severe, uncontrolled bacterial, fungal or viral infections (Active hepatitis B or C, history of HIV infection)
4. Pre-existing significant neurological disorder.
5. Active significant acute graft versus host disease (GVHD) or moderate/severe chronic GVHD requiring systemic steroids or other immunosuppressants within 4 weeks of enrolment.
6. Pregnant or lactating female.
7. The patient did not agree to use effective contraception during the treatment period and for the following 1 year.
8. A history of other malignant tumors.
9. Receiving systemic steroids therapy exceeding the equivalent of 0.5 mg/ kg/day of methylprednisolone, in the 7 days prior to CAR T-cell infusion
10. Receiving systemic immunosuppressive therapy in the 14 days prior to CAR T-cell infusion
11. Receiving intrathecal chemotherapy in the 7 days prior to CAR T-cell infusion

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Dose-limiting Toxicities (DLT) of CD19 CAR-T cells | Within 30 days after the last dose of CD19 CAR-T cells
  Patients will be continually assessed for unexpected adverse events using the NCI CTCAE (version 5.0) or unexpected early mortality 30 days post-infusion.
  The primary objectives for the Phase I study portion are to determine the maximum tolerated dose (MTD) and characterize the safety profile and dose-limiting toxicities (DLTs) of treatment with CD19 CAR-T cells in pediatric, adolescent and young adult patient's ≤ 25 years of age, with relapsed/refractory CD19+ ALL.

SECONDARY OUTCOMES:
Number of patients who achieve complete morphological remission | Within 30 days post CD19 CAR-T cells
  Number of patients who achieve complete morphological remission (Complete Response (CR) or Complete Response with Incomplete count recovery (CRi) in the bone marrow)

CONTACTS AND LOCATIONS:
Overall Officials: Tahereh Rostami, M.D, Principal Investigator — Research Institute for Oncology- Hematology and Cell Therapy (RIOHCT), Tehran University of Medical Sciences, Tehran, Iran; Naser Ahmadbeigi, PhD, Study Director — Gene Therapy Research Center, Shariati hospital, Tehran University of Medical Sciences, Tehran, Iran
Locations (2):
- Iran (2):
  - Gene therapy research center, Shariati hospital, Tehran university of medical sciences, Iran, Tehran
  - Research Institute for Oncology- Hematology and Cell Therapy (RIOHCT), Tehran University of Medical Sciences, Tehran

IPD SHARING:
Plan to Share IPD: Undecided